CLINICAL TRIAL: NCT07095257
Title: A Multicenter, Randomized, Double-blind, Positive Controlled, Phase III Trial to Evaluate the Safety and Efficacy of ZX-7101A for Oral Suspension in Pediatric Participants Aged 2 to 11 With Influenza
Brief Title: Study to Assess the Safety and Efficacy of ZX-7101A for Oral Suspension in Chinese Pediatric Participants 2 to 11 Years of Age With Influenza
Acronym: ZX-7101A-214
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZX-7101A-214
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Viral Infection
MeSH Terms: interventions — Suspensions; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZX-7101A for oral suspension (Experimental): A randomized phase III study with safety as primary endpoint was conducted in children (2-11 years old) with uncomplicated influenza. Eligible subjects were randomly assigned in a 2:1 ratio to receive either ZX-7101A for oral suspension （specification：10mg per bag）or oseltamivir phosphate for oral suspension （specification：0.36 g）.
  Preparation of suspension solution ZX-7101A: the specification of the dry suspension is 10 mg per bag. Add 10 ml of warm water for each bag, Mix well and take it all at once as soon as possible. Administer the dosage according to body weight.
  Interventions: Drug: ZX-7101A for oral suspension
- Oseltamivir phosphate for oral suspension (Active Comparator): A randomized phase III study with safety as primary endpoint was conducted in children (2-11 years old) with uncomplicated influenza. Eligible subjects were randomly assigned in a 2:1 ratio to receive either ZX-7101A for oral suspension （specification：10mg per bag）or oseltamivir phosphate for oral suspension （specification：0.36 g）.
  Administer the medication according to the weight specified in the label.
  Interventions: Drug: Oseltamivir phosphate for oral suspension

INTERVENTIONS:
Drug: ZX-7101A for oral suspension — ZX-7101A will be administered as oral suspension in a single dose on Day 1. Oseltamivir phosphate matching placebo will also be administered as oral suspension twice daily (BID) for 5 days.
  Arms: ZX-7101A for oral suspension
Drug: Oseltamivir phosphate for oral suspension — Oseltamivir phosphate will be administered as oral suspension BID for 5 days. Participants receiving oseltamivir will also receive ZX-7101A matching placebo as oral suspension, single dose on Day 1.
  Arms: Oseltamivir phosphate for oral suspension

SUMMARY:
The goal of this phase III study is to learn if ZX-7101A for oral suspension works to treat uncomplicated influenza in Pediatric Participants aged 2 to 11 years.

The main question it aims to answer is: What medical problems do participants have when taking drug ZX-7101A for oral suspension or Oseltamivir phosphate for oral suspension? Researchers will compare drug ZX-7101A for oral suspension to active comparator: Oseltamivir phosphate for oral suspension to see if drug ZX-7101A for oral suspension works to treat uncomplicated influenza in Pediatric Participants aged 2 to 11 years.

ELIGIBILITY:
Inclusion Criteria:

* ≥2 to<12 years of age at the time of randomization, males or females.
* Patients in the screening period met the following criteria:

  1. Rapid influenza diagnostic test (RIDT) or polymerase chain reaction (PCR) test positive;
  2. Axillary temperature ≥ 37.5℃ at screening; If taking antipyretics, axillary temperature ≥ 37.5℃ after taking the drug (more than 4 hours).
  3. At least one of the influenza-related respiratory symptoms is moderate or greater in severity: nasal congestion/runny nose and coughing.
* The first occurrence of influenza symptoms ≤ 48 hours from the time of patient randomization. The occurrence of symptoms is defined as:

  1. The body temperature first reached ≥ 37.5℃ (axillary/oral temperature) or 38.0℃ (rectal or tympanic temperature);
  2. Or the occurrence of at least one systemic or respiratory symptom: nasal congestion, sore throat, cough, muscle pain, headache, etc.
* The guardian of the participants must agree to participate in the study and sign a written informed consent form. For participants aged 8 years old and above, they must sign the informed consent form voluntarily (for participant under the age of 8, only the informed consent form signed by the guardian is required.); The participant s and/or their guardians agree to comply with all study procedures, including filling out the participant diary cards (the guardians of the subjects may assist in the assessment/filling).

Exclusion Criteria:

* Patients with severe or critically influenza virus infection (Meet any one of the following criteria).

  1. Severe cases with any of the following conditions： Dyspnea and/or increased respiratory rate: more than 30 breaths per minute for children over 5 years old; over 40 times per minute for children aged 2 to 5.

     Changes in consciousness: slow response, drowsiness, restlessness, convulsions, etc.

     Severe vomiting or diarrhea, with signs of dehydration. oliguria: Children with urine output<0.8 mL/(kg · h), or infants with daily urine output<200 mL/m2, preschool children<300 mL/m2, school aged children<400 mL/m2, or experiencing renal failure;
  2. Critical cases with any of the following conditions (Including but not limited to)： Respiratory failure; Acute necrotizing encephalomyopathy; Shock septic; Multiple organ dysfunction; Other serious clinical situations require intensive care Note: Refer to <the Expert Consensus on Diagnosis and Treatment of Childhood Influenza (2020 Edition)>
* High risk population for severe cases (meeting any of the following criteria):

  1. Accompanied by the following underlying diseases, and being clinically significant according to researchers' judgment, such as lung diseases (asthma, tracheopulmonary dysplasia, cystic fibrosis, etc.), liver diseases, kidney diseases, hematological diseases, heart diseases (congenital heart disease, chronic congestive heart failure [NYHA heart function classification III-IV], etc. But excluding hypertension without any other heart related symptoms), neurological and neuromuscular diseases that affect respiratory secretion clearance function (cognitive impairment, spinal cord injury, epileptic seizures, neuromuscular disorders, and cerebral palsy, etc), metabolic and endocrine system diseases.
  2. Immunocompromised individuals, such as patients with malignant tumors, organ or bone marrow transplants, HIV infections, or those who have been taking immunosuppressive drugs in the past 3 months.
  3. The electrocardiogram shows clinically significant QT corrected interval abnormalities (QTc ≥ 460ms) (QT corrected interval calculated according to Fridericia's formula, i.e. QTcF).
  4. Subjects require long-term use of aspirin or salicylate containing defined as those who need to take aspirin or salicylate containing drugs regularly per day for more than 14 days.
  5. With a body mass index (BMI) exceeding the criteria outlined in Appendix 2 of this protocol; During the screening period, patients with clinically significant bronchitis, pneumonia, pleural effusion, or interstitial lesions that identified by the researchers. If the researcher deems it necessary, imaging examinations (chest X-ray or chest CT) can be performed.
* Individuals who have experienced acute respiratory infections or otitis media and sinusitis within the past 2 weeks prior to screening.
* Combined with other respiratory infections, or requiring systemic anti infection treatment, or blood routine examination during screening with white blood cell count (WBC)>ULN (venous blood).
* Coughing up purulent phlegm or suffering from purulent tonsillitis.
* Have difficulty in swallowing medicine or have a history of gastrointestinal diseases that determined by researchers to seriously affect drug absorption.
* Suspected allergy to the active ingredients or excipients of the investigational drug.
* Have taken anti influenza virus drugs (including but not limited to: neuraminidase inhibitors, hemagglutinin inhibitors, M2 ion channel blockers, and cap structure dependent endonuclease (CEN) inhibitors, such as oseltamivir, zanamivir, paramivir, favipiravir, rimantadine, amantadine, abiidol, balosavir, etc.) within the past 7 days prior to screening.
* Received live or attenuated vaccines within the first 2 weeks of randomization or subjects who have received influenza vaccine within the first 2 weeks of randomization;
* Suspect or have a history of alcohol or drug abuse.
* Positive in pregnancy test.
* Participated in other clinical trials and used any other clinical trial drugs or devices within the 30 days prior to screening;
* Determined by the researchers to be unsuitable for participation in this clinical study.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From day1 up to day15
  The Number of Participants with Treatment-Related Adverse Event will be evalated as the change of vital signs, electrocardiogram, physical examination, and Laboratory test compared with the baseline.

SECONDARY OUTCOMES:
Time to Alleviation of Influenza Signs and Symptoms | From day1 up to day15
  Time to alleviation of influenza signs and symptoms is defined as the length of time taken from the start of treatment to the point at which all of the following criteria are met (Standard a or b) and remain so for at least 21.5 hours:
  1. Body temperature returns to normal (axillary temperature ≤ 37.2℃)
  2. In the CARIFS scale, a score of 0 (no problem) or 1 (minor problem) for cough ,rhinobyon or nasal symptoms.
Duration of fever | From day1 up to day15
  Length of time taken by participants to return to afebrile state [axillary temperature ≤ 37.2°C] and remaining so for at least 21.5 hours.
Time to Alleviation of Symptoms | From day1 up to day15
  Symptom recovery time: Defined as the period from the start of the study treatment until all 16 assessment items in the CARIFS were evaluated as being asymptomatic or mild, and remained so for at least 21.5 hours.
Time to Return to Normal Health and Activity | From day1 up to day15
  Time to Return to Normal Health and Activity
The time influenza RNA turns negative | From day1 up to day15
  Defined as the time from initiation of treatment until the first influenza viral RNA falls below the lower limit of quantification (measured by RT-PCR)
The time Virus Titer turns negative | From day1 up to day15
  Defined as the time from initiation of treatment until the first viral titer falls below the lower limit of quantification
Change From Baseline in the Amount of Virus RNA (RT-PCR) and Influenza Virus Titer at each visit | Baseline, Day 2,3,5,9,15
  Change From Baseline in the Amount of Virus RNA (RT-PCR, unit: log10virus particles/mL) and Influenza Virus Titer (unit: log10TCID50/ML) at each visit
Percentage of Participants With Positive Influenza Virus Titer at each visit (measured by RT-PCR) | Baseline, Day 2,3,5,9,15
  Percentage of Participants With Positive Influenza Virus Titer at each visit (measured by RT-PCR)(unit: %)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No